CLINICAL TRIAL: NCT03310177
Title: Compartmental Analysis of Metabolite Profiles Associated With Disease Phenotype in Smokers With and Without Chronic Obstructive Pulmonary Disease
Brief Title: Relationship Between Metabolic Profile and Clinical Phenotype in Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Bei He, Professor and Chief in Department of Respiratory Medicine, Peking University Third Hospital
Other Study IDs: Metabolomcs-HB
Record Dates: First submitted 2017-10-10; First posted 2017-10-16 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Metabolomics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD: The smokers who are diagnosed as chronic obstructive pulmonary disease according to GOLD guideline.
- healthy control: The healthy controls without chronic obstructive pulmonary disease

SUMMARY:
Despite the high prevalence of chronic obstructive pulmonary disease (COPD), there continues to be a large gap in our understanding of disease pathogenesis and mechanisms accounting for large variability in disease phenotype. Untargeted metabolomics is an ideal approach to uncover the metabolic basis of disease, as well as discover unique drug target opportunities aimed at these nodal metabolic drivers of disease. There are very limited data from metabolomics studies from plasma/serum and exhaled breath condensate that suggest certain metabolic pathways or metabolites might predict the presence and/or severity of COPD phenotypes.

Here, the investigators hope to generate comprehensive, compartment specific (blood and lung) metabolite profiles that will be correlated with various clinical phenotypes of COPD, using a complementary approach of untargeted nuclear magnetic resonance (NMR) and liquid chromatography (LC)- mass spectroscopy (MS) -based metabolomics.

DETAILED DESCRIPTION:
Despite the high prevalence of chronic obstructive pulmonary disease (COPD), there continues to be a large gap in our understanding of disease pathogenesis and mechanisms accounting for large variability in disease phenotype. Untargeted metabolomics is an ideal approach to uncover the metabolic basis of disease, as well as discover unique drug target opportunities aimed at these nodal metabolic drivers of disease. There are very limited data from metabolomics studies from plasma/serum and exhaled breath condensate that suggest certain metabolic pathways or metabolites might predict the presence and/or severity of COPD phenotypes.

The investigators hypothesize that: 1) smokers with COPD will have a metabolomics signature that is distinct from healthy non-COPD smokers; 2) this signature will be associated with clinically relevant manifestations of disease (e.g., GOLD classification, PFT).

The availability of biosamples from a well-characterized population of smokers with and without COPD, combined with our established in-house metabolomics expertise, will robustly allow to test these novel hypotheses. The investigators hope to generate comprehensive, compartment specific (blood and lung) metabolite profiles that will be correlated with various clinical phenotypes of COPD, using a complementary approach of untargeted nuclear magnetic resonance (NMR) and liquid chromatography (LC)- mass spectroscopy (MS) -based metabolomics. Moreover, this strategy may identify previously unrecognized metabolic pathways that are dysregulated in COPD. Collectively, these data will be used to direct a prospective clinical study to determine the association between metabolomics signatures and clinical outcomes.

ELIGIBILITY:
IInclusion Criteria:

1. males aged 40-80;
2. diagnosed with COPD according to the GOLD guidelines;
3. clinically stable patients without medication changes or exacerbation in two months;
4. smoking history of more than 10 pack years

Exclusion Criteria:

1. diagnosed with unstable cardiovascular diseases, significant renal or hepatic dysfunction or mental incompetence;
2. diagnosed with asthma, active pulmonary tuberculosis, diffuse panbronchiolitis, cystic fibrosis, clinically significant bronchiectasis, exacerbation of COPD or pneumonia in two months;
3. prescribed immunosuppressive medications.

Ages: 40 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Clinically stable patients with COPD and controls without COPD are enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2015-12-10 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Metabolites that can predict the progress of lung function | 3 months
  The study is aimed to investigate the relationship between the metabolites and the progress of lung function in COPD

SECONDARY OUTCOMES:
Metabolites that can predict the severity of emphysema | 3 months
  The association between metabolites and emphysema is also investigated
Metabolites that are associated with inflammatory mediators | 3 months
  The association between metabolites and inflammatory mediators is also investigated

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Diao W, Labaki WW, Han MK, Yeomans L, Sun Y, Smiley Z, Kim JH, McHugh C, Xiang P, Shen N, Sun X, Guo C, Lu M, Standiford TJ, He B, Stringer KA. Disruption of histidine and energy homeostasis in chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2019 Sep 3;14:2015-2025. doi: 10.2147/COPD.S210598. eCollection 2019. PMID 31564849